CLINICAL TRIAL: NCT06774131
Title: A Phase 3, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of UGN-104, a Novel Formulation of UGN-101, for the Treatment of Patients With Low-grade Upper Tract Urothelial Cancer (LG-UTUC)
Brief Title: A Phase 3 Single-arm Study of UGN-104 for the Treatment of Low-grade Upper Tract Urothelial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UT002; 2024-519343-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma; Urothelial Carcinoma
Keywords: UTUC; Low Grade UTUC; Low-grade Upper Tract Urothelial Cancer; UGN-104; Mitomycin; Nephrostomy Tube; LG-UTUC; UGN-101
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UGN-104 (Experimental): Patients will receive UGN-104 once weekly for 6 weeks (a total of 6 doses). The dose of UGN-104 to be instilled is 4 mg mitomycin per 1 mL sterile hydrogel via ureteral catheter (retrograde administration) or nephrostomy tube (antegrade administration).
  Patients who have a CR at the PDE Visit will enter the Follow-up Period and may receive UGN-104 as maintenance treatment once monthly for 11 months (a total of 11 doses) at the discretion of the investigator.
  Interventions: Drug: UGN-104

INTERVENTIONS:
Drug: UGN-104 — UGN-104 consists of mitomycin and sterile hydrogel (a proprietary thermally responsive gel) that is used to reconstitute mitomycin before instillation. The reverse thermal properties of UGN-104 allow for local administration of mitomycin as a liquid under chilled conditions, with subsequent conversion to a semi-solid gel depot following instillation into the UUT.
  Other Names: UGN-104 (mitomycin) for pyelocalyceal solution

SUMMARY:
This study will evaluate the efficacy and safety of UGN-104, a new formulation of UGN-101 (approved in the United States and Israel as JELMYTO [mitomycin] for pyelocalyceal solution), instilled in the upper urinary tract (UUT) of patients with low-grade upper tract urothelial cancer (LG-UTUC).

DETAILED DESCRIPTION:
Eligible patients will be treated with UGN-104 once weekly for 6 weeks (a total of 6 doses).

Efficacy will be assessed by the complete response rate (CRR) at the Primary Disease Evaluation (PDE) Visit (approximately 3 months after the first instillation). Response will be determined based on central laboratory interpretation of UUT wash urine cytology and visual evaluation (ureteroscopy). Biopsy of any remaining or new lesions will be performed where technically feasible and the central laboratory histopathology assessment will also be used in the response determination, if applicable.

Patients who have a complete response (CR) at the PDE Visit, defined as having no detectable disease (NDD), will enter the Follow-up Period of the study. During the Follow-up Period, patients may receive UGN-104 as maintenance treatment at the discretion of the investigator. The maintenance regimen is once monthly for 11 months (a total of 11 doses) and should start as soon as possible (no longer than 3 weeks) after CR is determined at the PDE Visit.

All patients in the Follow-up Period, regardless of whether they receive maintenance treatment, will return to the clinic every 3 months for evaluation of response and will remain on study for 12 months after the PDE Visit or until disease recurrence, disease progression, or death, whichever occurs first.

Patients who have a non-complete response (NCR) at the PDE Visit will be considered to have completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and protocol.
2. Naive or recurrent patients with LG, non-invasive UTUC in the pyelocalyceal system, with the following disease characteristics:

   1. At least 1 measurable papillary LG tumor, evaluated visually, ≤ 15 mm. The largest lesion should not exceed 15 mm. Debulking to ≤ 15 mm is permitted.
   2. Biopsy taken from at least 1 tumor located above the ureteropelvic junction revealing LG urothelial carcinoma (UC). Patients who have been biopsied within 8 weeks before Screening for this study and shown to have LG UC may have these historical biopsies used for enrollment into the study and do not require repeat biopsy during Screening.
   3. Patient should have at least 1 remaining papillary LG tumor evaluated visually with a diameter of at least 5 mm post-biopsy.
   4. Wash urine cytology sampled from the pyelocalyceal system documenting the absence of high-grade (HG) UC, diagnosed not more than 8 weeks before Screening.
   5. Patients with bilateral LG-UTUC may be enrolled if at least 1 side meets the inclusion criteria for the study and if the other kidney does not require further treatments. (The disease in the other kidney must be completely ablated before receiving treatment in the study.) Note: If both upper tracts meet inclusion criteria, the treating urologist in consultation with the sponsor's medical monitor can decide which side to treat in the study. The pyelocalyceal system not under study must be free of cancer before the first instillation on the side to be treated in the study.
3. Patients with Eastern Cooperative Oncology Group (ECOG) performance status < 3 (with Karnofsky > 40).
4. Patients with life expectancy > 24 months at time of Screening.
5. Patients must have adequate organ and bone marrow function as determined by the following routine laboratory tests:

   1. Leukocytes ≥ 3,000/μL (≥ 3 × 10^9/L).
   2. Absolute neutrophil count ≥ 1,500/μL (≥ 1.5 × 10^9/L).
   3. Platelets ≥ 100,000/μL (≥ 100 × 10^9/L).
   4. Hemoglobin ≥ 9.0 g/dL.
   5. Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN.
   7. Alkaline phosphatase ≤ 2.5 × ULN.
   8. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min.
6. Patient has no active urinary tract infection (UTI) as confirmed by urine culture or urinalysis. Note: In case of a symptomatic UTI the patient will be treated with antibiotics and the instillation will be postponed until resolution. In the case of asymptomatic bacteriuria, the use of prophylactic antibiotics and postponement of treatment is at the discretion of the investigator.
7. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for clinical study participants.

Female patients of childbearing potential (defined as premenopausal women who have not been sterilized) and male patients with female partners of childbearing potential must agree to use 2 acceptable forms of effective contraception from enrollment through 6 months post treatment. Sexually active male patients must agree to use a condom during intercourse for at least 48 hours after each instillation.

Acceptable methods of birth control considered to have a low failure rate (ie, less than 1% per year) when used consistently and correctly include implants, injectable, combined (estrogen/progesterone) oral contraceptives, intrauterine devices (only hormonal), condoms with spermicide, sexual abstinence* or vasectomized partner.

* Sexual abstinence is defined as refraining from intercourse from enrollment through 6 months post treatment. Periodic abstinence (calendar, symptothermal, post-ovulation methods) is NOT an acceptable method of contraception.

Exclusion Criteria:

1. UC specific exclusions:

   1. Patient received Bacillus Calmette-Guérin (BCG) treatment for UC during the 6 months before enrollment.
   2. The patient has untreated concurrent UC in locations other than the target area (unless treated and resolved during Screening); ie, ureteral and lower urinary tract tumors must be completely ablated before entry.
   3. Patient has a history of carcinoma in situ (CIS) in the urinary tract.
   4. Patient has a history of invasive UC in the past 5 years.
   5. Patient has a history of HG papillary UC in the urinary tract in the past 2 years.
2. Patient is actively being treated or intends to be treated with systemic chemotherapy during the duration of the study.
3. Any other malignancy diagnosed within 2 years before enrollment with the exception of:

   1. Basal or squamous cell skin cancers.
   2. Noninvasive cancer of the cervix.
   3. Any other cancer deemed to be of low risk for progression or patient morbidity during the study period in the opinion of the investigator.
4. Patient with urinary obstruction such that there is an inability to deliver the study treatment to the pyelocalyceal system either via ureteral catheter (retrograde administration) or nephrostomy tube (antegrade administration).
5. Known allergy or sensitivity to any component of the study treatment (including excipients) that in the investigator's opinion cannot be readily managed.
6. Patient has an intractable bleeding disorder (eg, coagulation factors deficiencies, Von Willebrand disease).
7. Patient is currently receiving any other investigational product, has participated in a research protocol involving administration of an investigational product in the past 30 days, or plans to participate in a research protocol involving administration of an investigational product during study conduct.
8. Patient was previously treated with JELMYTO (product code UGN-101) for UTUC.
9. Women who are pregnant (positive urine or serum pregnancy test), planning to become pregnant during the study period, or who are breastfeeding are not eligible to enroll.
10. Patient has any other medical or mental condition(s) that make(s) his/her participation in the study unadvisable in the opinion of the investigator.
11. Where applicable per country regulation, the patient must not be currently committed to an institution by virtue of an order issued by either judicial or administrative authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | 3 months
  CRR is defined as the proportion of patients who achieved CR at the PDE Visit.

SECONDARY OUTCOMES:
Duration of response (DOR) | 12 months
  DOR is defined as the time from the date of evidence of CR at the PDE Visit to the earliest date of recurrence, progression, or death due to any cause, whichever occurred first.
Durable complete response (DCR) rate | 12 months
  DCR rate at scheduled disease assessment time points, defined as the proportion of patients who achieved CR at the PDE Visit and maintained CR (ie, no detectable disease) up to that particular follow-up disease assessment.
Incidence of treatment-emergent adverse events (TEAEs), serious TEAEs, TEAEs of special interest, and abnormal clinical laboratory test results (hematology and serum chemistry) | 15 months
  The number of patients with each type of event will be summarized.
Mitomycin plasma concentrations | 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-104
  Mitomycin plasma concentrations will be assessed in a subset of patients treated with UGN-104.
Mitomycin maximum plasma concentration (Cmax) | 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-104
  Mitomycin Cmax will be assessed in a subset of patients treated with UGN-104.
Mitomycin time to maximum plasma concentration (tmax) | 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-104
  Mitomycin tmax will be assessed in a subset of patients treated with UGN-104.
Mitomycin area under the concentration-time curve (AUC) | 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-104
  Mitomycin AUC will be assessed in a subset of patients treated with UGN-104.
Mitomycin terminal half-life (t1/2) | 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-104
  Mitomycin t1/2 will be assessed in a subset of patients treated with UGN-104.

CONTACTS AND LOCATIONS:
Overall Officials: Derrick McKinley, MD, Study Director — UroGen Pharma
Locations (41):
- United States (18):
  - Urology Centers of Alabama, Homewood, Alabama
  - Arizona State Urological Research Institute, LLC ("ASURI"), Chandler, Arizona
  - Michael G Oefelein Clinical Trials, Bakersfield, California
  - University of California, Irvine, Orange, California
  - BioResearch Partners Aventura, Aventura, Florida
  - UF Health Cancer Center University of Florida, Gainesville, Florida
  - BioResearch Partners Hialeah, Hialeah, Florida
  - Urology Center of Iowa Research, Clive, Iowa
  - The Urology Center, P.C., Omaha, Nebraska
  - University of Cincinnati Medical Center (UCMC), Cincinnati, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Carolina Urologic Research Center, LLC, Myrtle Beach, South Carolina
  - Low county Urology Clinics, North Charleston, South Carolina
  - Amarillo Urology Research, Amarillo, Texas
  - UPNT Research Institute, LLC, Arlington, Texas
  - Texas Urology Specialists-Austin, Austin, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
- Bulgaria (2):
  - MHAT Haskovo AD, Haskovo
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov," Sofia, Clinic of Urology, Sofia
- Georgia (4):
  - LTD "Israel-Georgian Medical Research Clinic "Healthycore", Tbilisi
  - JSC "Vian"-I.Bokeria University Hospital, Tbilisi
  - LTD "Geo Hospitals", Tbilisi
  - LTD "Tbilisi State Medical University and Ingorokva High Medical Technology University Clinic", Tbilisi
- Israel (5):
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Department of Urology, Kefar Sava
  - Rabin Medical Center - Hasharon hospital, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Assaf Harofeh hospital, Shamir Medical Center, Ẕerifin
- Poland (3):
  - IN-VIVO Limited Liability Company, Bydgoszcz
  - NZOZ Silesian Urology Hospital, Katowice
  - Jan Mikulicz-Radecki University Clinical Hospital in Wroclaw, Wroclaw
- Romania (4):
  - Municipal Clinical Hospital Cluj-Napoca, Cluj-Napoca
  - Regional Institute of Oncology Iasi, Iași
  - Bihor County Emergency Clinical Hospital, Oradea
  - Timisoara County Clinical Emergency Hospital Pius Brinzeu, Timișoara
- Spain (5):
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia